CLINICAL TRIAL: NCT04665141
Title: Similarities and Differences of Biological Therapies for Severe Asthma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Regional de Malaga (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-ALER-2021-01
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab; Omalizumab; reslizumab; benralizumab; dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of care: Patients with severe asthma being treated with non-biological standard therapies, mainly systemic corticosteroids.
- Biological therapies: Patients with severe asthma being treated with omalizumab, mepolizumab, reslizumab, benralizumab, or dupilumab.
  Interventions: Biological: Mepolizumab; Biological: Omalizumab; Biological: Reslizumab; Biological: Benralizumab; Biological: Dupilumab

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab will be prescribed freely by the treating physician according to real-life conditions.
  Other Names: Nucala®
  Groups: Biological therapies
Biological: Omalizumab — Omalizumab will be prescribed freely by the treating physician according to real-life conditions.
  Other Names: Xolair®
  Groups: Biological therapies
Biological: Reslizumab — Reslizumab will be prescribed freely by the treating physician according to real-life conditions.
  Other Names: Cinqair®
  Groups: Biological therapies
Biological: Benralizumab — Benralizumab will be prescribed freely by the treating physician according to real-life conditions.
  Other Names: Fasenra®
  Groups: Biological therapies
Biological: Dupilumab — Dupilumab will be prescribed freely by the treating physician according to real-life conditions.
  Other Names: Dupixent®
  Groups: Biological therapies

SUMMARY:
This is an ambispective multicenter longitudinal observational study to evaluate the efficacy and safety profile of biological therapies in patients diagnosed with severe asthma in real life conditions.

DETAILED DESCRIPTION:
The use of biologicals to treat severe asthma has been implemented in a regular basis while information on long term effectiveness and safety is lacking. It is necessary to establish strategies to closely monitor the possible occurrence of reactions, adverse effects of innovative biological medicines used to treat severe asthma.

In this study the investigators want to evaluate the comparative effectiveness, utilization patterns, long-term safety, and use in special groups in real-life conditions in severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any age: adults and children.
* Diagnosis of severe asthma as given by the treating physician, and defined as an asthma that remains uncontrolled in despite adherence with maximal optimized therapy and treatment of contributed factors, or asthma that worsens when high dose treatment is decreased.
* Being treated or not (control group) with biological drugs.
* Signed Informed Consent.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients, adults and children, with a diagnosis of severe asthma in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Treatment dose scheduling and changes of dose throughout the study. | 2 years after inclusion
Number of treatment discontinuations and causes of interruption throughout the study. | 2 years after inclusion
Incidence of Relevant Treatment-Related Adverse Events recorded throughout the study. | 2 years after inclusion
Severity of Treatment-Related Adverse Events recorded throughout the study. | 2 years after inclusion
Change of asthma control during the treatment. | 2 years after inclusion
  Number of asthma exacerbations, change in FEV1, ACT, and blood eosinophilia, need of add-on medication, inhaled medication and systemic corticosteroids.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil-Hospital Regional Universitario de Málaga, Málaga, Spain